CLINICAL TRIAL: NCT00338364
Title: Painful Procedures in the Emergency Department:Does a Formal Program in Distracting Techniques for Parents and Children Reduce Pain and Anxiety in Children?
Brief Title: Painful Procedures in the Emergency Department: A Distraction Intervention
Acronym: ERPain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: Mayday Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3202; Mayday grant
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Pediatric Pain and Anxiety
Keywords: Pediatric pain; Pediatric anxiety; Painful procedures
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 50% randomized to receive distraction during painful procedure
  Interventions: Behavioral: PAT
- Control (No Intervention): 50% randomized to receive no distraction during painful procedure

INTERVENTIONS:
Behavioral: PAT — Coping and Distraction Intervention
  Arms: Treatment

SUMMARY:
This study is designed to assess the effectiveness of the video-based intervention over and above current standard practice for pain control in the pediatric emergency department (ED). This is a single-center trial based at the IWK Health Centre. The primary outcome will be based on the CAMPIS coding of the video-taped pain response of the research participants.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the pain and anxiety that children experience when they have venipuncture procedures performed can be reduced by a video-based distraction and coping strategy intervention. An instructional video has been designed to educate parents and children about what is going to happen during the venipuncture procedure; to teach coping skills that can be used before and during the painful procedure; and to provide distraction during the procedure by using an entertaining video segment.

Approximately 168 children (6-12 years of age)who are seen in the IWK ED requiring venipunctures for blood collection or IV starts will be randomized. PArent and child training in distraction and coping strategies will be provided by means of a self-administered video-delivery via a portable DVD player. Fifty percent of the eligible participants will receive the distraction and coping strategies intervention and 50% will receive the standard medical care provided by the IWK ED. Those receiving standard care will be evaluated for outcome results and then be compared to the intervention group. It is expected that children who receive the intervention will report less pain and anxiety associated with venipunctures than those who receive standard care.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible for this study if they:

* are between 6-12 years of age
* are presenting in the IWK Emergency Department who require a venipuncture for blood collection or IV initiation.
* are able to read and speak english
* provide written parental authorization and verbal child assent

Exclusion Criteria:

Participants will be excluded for this study if they:

* are in critical condition as determined by ED staff
* are in significant pain for other reasons other than the venipuncture
* have severe cognitive delay
* who require sedation for the venipuncture as determined by the ED staff

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 189 (Actual)
Dates: Start 2006-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
CAMPIS coding of visual pain response video-recorded during the procedure | continuous

SECONDARY OUTCOMES:
Child pain ratings (Faces Pain Scale Revised) | post procedure
Child anxiety ratings | post procedure
CHEOPS analysis | post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. McGrath, PhD., Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada